CLINICAL TRIAL: NCT02656992
Title: Effects of High Intensity Inspiratory Muscle Training on Exercise Capacity in Patients With Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozge OZER, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 13/292
Record Dates: First submitted 2015-11-20; First posted 2016-01-15 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; High-intensity inspiratory muscle training
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-IMT group (Experimental): Intervention group receive supervised training sessions three times per week for 8 weeks. Each sessions lasted 21 minutes and comprised seven cycles of 2 minutes of breathing on an inspiratory threshold device followed by 1 minute of rest. High-IMT was performed at the maximal load tolerable for each 2-minute work interval and was progressively increased over the training period.
  Interventions: Device: Inspiratory muscle training group
- Control group (Sham Comparator): Control group was prescribed at 10% of baseline maximal inspiratory pressure, and remained at this level during all training sessions for 8 weeks.
  Interventions: Device: Inspiratory muscle training group

INTERVENTIONS:
Device: Inspiratory muscle training group

SUMMARY:
Reduced exercise tolerance is commonly reported in patients with bronchiectasis. The purpose of this study is to evaluate the effects of high-intensity inspiratory muscle training (High-IMT) and sham High-IMT (control) on exercise capacity, respiratory muscle function (strength and endurance) and health related quality of life in patients with bronchiectasis.

DETAILED DESCRIPTION:
Bronchiectasis often demonstrates decreased exercise tolerance, marked dyspnea and fatigue. The causes are multifactorial and include altered pulmonary mechanics, inefficient gas exchange, decreased muscle mass, and psychological status, which all lead to a progressive detraining effect. Essentially both the pathology and the functional manifestations of bronchiectasis increase the demand for inspiratory muscle work and that contribute to dyspnea and exercise limitation.

In recent studies reduced strength of respiratory muscles are investigated in bronchiectasis and can be contribute the exercise limitation. Additionally IMT has shown to improve respiratory muscle function, exercise tolerance and dyspnea in patients with bronchiectasis. Despite this, the number of studies are inadequate and so the optimal training protocol remains still to be defined. In this study the researchers want to investigate the effects of high-intensity inspiratory muscle training in functional results in patients with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bronchiectasis with high resolution computed tomography
* being 18-65 years of age
* being able to walk and co-operate

Exclusion Criteria:

* acute exacerbation or change in drugs or usage of antibiotics in last 3 weeks
* neurological disease, severe orthopaedic problem or advanced heart failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2017-12-25 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Exercise capacity using incremental shuttle walk test and 6-minute walk test | Baseline to 8 weeks
  * The incremental shuttle walk test will be performed in an enclosed corridor. Patients are required to walk back and forth, turning around two cones placed 9 meters apart making the shuttle distance 10 meters long. Patients will follow the rhythm dictated by the audio signal.
  * 6-minute walk test will be performed in a long, straight, enclosed corridor 30 meters in length. Patients are required to walk in their walking speed with standardised instructions. The distance walked by subjects during 6 minutes will be recorded.

SECONDARY OUTCOMES:
Respiratory muscle strength | Baseline to 8 weeks
  Respiratory muscle strength is measured through maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) using a handheld device.
Respiratory muscle endurance | Baseline to 8 weeks
  Respiratory muscle endurance is assessed with constant and progressive loading protocols which subjects breathe against threshold loads.
Health related quality of life is assessed with Leicester Cough Questionnaire | Baseline to 8 weeks
Dyspnea severity is assessed with The Modified Medical Research Council Dyspnea Scale (MMRC) | Baseline to 8 weeks
Fatigue severity is assessed with Fatigue Severity Index | Baseline to 8 weeks
Severity of disease is assessed with Bronchiectasis Severity Index | Baseline to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ozge Ozer, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozalp O, Inal-Ince D, Cakmak A, Calik-Kutukcu E, Saglam M, Savci S, Vardar-Yagli N, Arikan H, Karakaya J, Coplu L. High-intensity inspiratory muscle training in bronchiectasis: A randomized controlled trial. Respirology. 2019 Mar;24(3):246-253. doi: 10.1111/resp.13397. Epub 2018 Sep 12. PMID 30209855